CLINICAL TRIAL: NCT06299917
Title: WORK-ON - Vocational Rehabilitation for People with Chronic Inflammatory Arthritis - a Randomised Controlled Trial
Brief Title: WORK-ON Vocational Rehabilitation for People with Inflammatory Arthritis
Acronym: WORK-ON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Center for Expertise in Rheumatology (Other)
Collaborators: Odense Patient Data Explorative Network (Other); The Danish Rheumatism Association (Other); Danish Association of Occupational Therapist (Other); Schaufuss foundation (Unknown)
Responsible Party: Principal Investigator, Jette Primdahl, Professor in rheumatology rehabilitation, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CeViG; S-20232000 - 3 (Other: Committees on Health Research Ethics for Southern Denmark)
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Axial Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Single center parallel randomized study
Masking Description: Statistical analyses will be blinded for group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WORK-ON (Experimental): The 6-months WORK-ON VR includes three parts in addition to usual care:
  1: A coordinating occupational therapist (OT) (10 hours): An initial assessment and goal setting process. Support to navigate offers in the municipalities and to involve the employer.
  Provides individual support in relation to the goals agreed upon. After six months, goals, the patients' progress during the intervention and future need for support are evaluated.
  Follow-up consultation 12 months after baseline. Group sessions to meet with others in the same situation and exchange experiences.
  1. Legislative offers (social worker and coordinating OT)
  2. Acceptance of the disease in relation to work (nurse and the coordinating OT).
  3. Coping strategies (physiotherapist and coordinating OT).
  4. Follow-up (nurse and the coordinating OT). Up to 8 individual consultations are offered with a physiotherapist, nurse and or social worker to achieve the goals.
  Interventions: Other: WORK-ON
- Usual care (No Intervention): Both the intervention and the control group will receive usual care in the outpatient department. Usual care consists of planned outpatient consultations every 3-12 months depending on the patient's needs, alternating between a rheumatologist and rheumatology nurses. In addition, they have access to support from a telephone help-line to the rheumatology nurses. The planned consultations include review of blood tests, joint examinations, review of completed questionnaires in DANBIO, which is a national rheumatology quality database, adherence to the pharmacological treatment and evaluation of whether pharmacological adjustment is necessary. The nurses can provide limited occasional patient education tailored to the specific patient on management of their disease, medications and symptoms. The participants in the control group will be offered pamphlets for their employer and colleagues (Dear Employer and Dear colleague)

INTERVENTIONS:
Other: WORK-ON — The intervention includes three parts: 1) a coordinating occupational therapist, 2) four group sessions and 3) Individual consultations based on the agreed upon goals.
  Arms: WORK-ON

SUMMARY:
People with chronic inflammatory arthritis (IA) (rheumatoid arthritis, axial spondyloarthritis, and psoriatic arthritis), often have a reduced work ability. Up to 40% lose their job in the first years after diagnosis. Consequently, they are at high risk of losing their jobs and being permanently excluded from the labour market. Therefore, a new context-specific vocational rehabilitation (VR) for people with IA was developed, based on the Medical Research Council's framework for complex interventions. The 6-months VR is called WORK-ON and consists of three parts: 1) a coordinating occupational therapist who performs an initial assessment and goalsetting process and supports cooperation between relevant partners and navigation between sectors, 2) Four group sessions with peers and if needed, 3) Individual sessions with a social worker, nurse, or physiotherapist. The objective of the WORK-ON trial is to test the overall efficacy on work ability compared to a control group who receives usual care and pamphlets for their employer and colleagues.

Based on the experiences from a feasibility study, WORK-ON will be conducted as a randomised controlled trial. Patients with IA, aged 18 years or older, experiencing job insecurity will be randomised to one of two groups: the WORK-ON VR group or usual care (control group). The primary outcome; work ability measured is measured by Work Ability Index single item, at baseline, 6, 12, 18 and 30 months after baseline. Secondary outcomes are absenteeism, presenteeism, overall work impairment, activity impairment, job loss, quality of life, mental well-being, fatigue, sleep, physical activity, occupational balance and pain. Secondary outcomes are measured at baseline, 6 and 12 months after baseline. In addition, work ability, working hours per week and job loss are measured at 18 and 30 months after baseline.

DETAILED DESCRIPTION:
In Denmark, about 100,000 people are diagnosed with chronic autoimmune inflammatory arthritis (IA). In this study, IA includes rheumatoid arthritis (RA), axial spondyloarthritis (axSpA), and psoriatic arthritis (PsA). Despite major advances in pharmacological treatment, there are still unmet needs among people with IA. Many experience pain, fatigue, sleep problems, anxiety, physical disability and/or problems with participation in everyday activities, including paid work.

Up to 40% lose their job in the first years after being diagnosed. Support to maintain work needs to be offered early, as it is difficult to get back to work if long-term absenteeism occurs. In 2013, people with RA had 5.6 more days away from work due to sickness absenteeism than people without RA in Denmark. This corresponds to more than 50,000 days of sickness absenteeism per year and a productivity loss of 67.3 million DKK (app. 9 million EURO).

Being able to work is of great importance to the experience of identity and quality of life among people with RA. People with IA struggle to find a balance between their disease, paid work, and other aspects of everyday life. In a systematic review on interventions to prevent job loss among people with IA, showed that strategies such as job accommodation, job coaching, physical exercise, and ergonomic and vocational counselling may have an effect on job loss, work ability and absenteeism. The study pointed to a need for a context specific tailored vocational rehabilitation (VR). Given that VR depends on the context, and countries have different social security systems, it is important to develop and test a context-specific VR.

At the Danish Hospital for Rheumatic Diseases (DHR), a VR called 'WORK-ON' for people with IA who consider they are at risk of job loss within the following two years was developed based on the updated Medical Research Counsil's framework for developing and evaluating Complex Interventions. In the development of WORK-ON, relevant stakeholders including patient research partners were involved. In addition, a logic model to help explain the associations between resources and outcomes of the intervention was developed.

In 2022-2023 the feasibility of the WORK-ON VR was tested in 19 participants. Based on the results from the feasibility test, the WORK-ON VR was slightly adjusted based on qualitative evaluations with patients and rehabilitation clinicians.

Work ability is considered to be a proxy for future job loss.

Aim: To test the efficacy of the adjusted WORK-ON VR on work ability relative to usual care.

Material and Methods: This study was developed in accordance with the Usual Protocol Items: Recommendations for Interventional Trials (SPIRIT) reporting guideline. The trial is planned as a randomised controlled trial (RCT) with a two group parallel design. Participants will be allocated 1:1 to either the WORK-ON VR (the intervention group) or usual care (the control group) stratified by diagnosis and disease duration.

The trial is based on a two-sided superiority framework where the primary null hypothesis is that there is no difference between the groups (H0: µ[I] = µ[C]) on change in the primary outcome.

Study setting: The WORK-ON VR will be carried out at the DHR, which is a specialised hospital for rheumatic diseases and rehabilitation owned by the patient organisation, the Danish Rheumatism Association. The hospital has a large outpatient department and offers inpatient rehabilitation for patients with rheumatic diseases from all five regions in Denmark.

Recruitment: Before each outpatient consultation at the DHR, all patients with IA complete questionnaires collected in the national rheumatology quality database, DANBIO at a touchscreen in the waiting area or at a mobile phone, tablet or computer at home. An initial screening will be performed in DANBIO. For patients with a diagnosis of RA, axSpA or PsA and 18 ≤ age ≤65, the regular questionnaires at the present visit are followed by a question whether the patient is in paid work or not. If yes, question #6 from the WAI questionnaire follows: "Do you believe, according to your present state of health, that you will be able to do your current job two years from now?". If the patient answers "unlikely" or "not certain", a short information about WORK-ON is shown as a pop-up text at the screen. If the patient is interested to hear more about the WORK-ON VR, they are prompted to insert their phone number. Interested patients are contacted by a project member by phone to offer more information about the study within the following week. If still interested, a project member will check the remaining in- and exclusion criteria in the patient's medical journal. If the patient fulfils all eligibility criteria, written participant information is sent by e-mail to allow interested patients time for consideration before they are asked to give their written consent. If the patient wants to participate, a written consent is collected through REDCap

Randomisation and blinding: Randomisation and data collection will be performed using the Research Electronic Data Capture (REDCap) hosted by the Open Patient data Explorative Network (OPEN). OPEN is a safe storage and analysis environment in the Region of Southern Denmark. REDCap is a secure web application to be used for randomisation and for building and managing online surveys. Randomisation will be performed using block randomisation and is stratified by diagnosis. Due to the nature of the intervention, neither the rehabilitation clinicians nor the participants can be blinded. The statistical analyses will be performed blinded to group allocation.

Ethics: The participants will be informed verbally and in writing about the study before providing their written consent to participate before the first consultation. The study will be conducted in accordance with the Helsinki Declaration. The leaflet," Research subjects' rights in health science research" published by the Danish National Committee on Health Research Ethics, is provided to all participants. The Regional Committees on Health Research Ethics waived the need for a formal approval (Journal number S-20232000-3). Data will be stored and managed in OPEN, which adheres to the European General Data Protection Regulations and the Danish data protection law.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years.
* Diagnosed with RA, PsA or axSpA by a rheumatologist.
* Undertakes paid work (full- or part-time work or studying).
* Able to read and understand Danish.
* Answers 'unlikely' or 'not certain' to question #6 from the WAI questionnaire: 'Do you believe, according to your present state of health, that you will be able to do your current job two years from now?' (36).
* Willing to participate in an RCT of the modified WORK-ON VR.

Exclusion Criteria:

* Planned or present adjustments of the pharmacological anti-rheumatic treatment (DMARDs, glucocorticoid) within the last three months.
* Presence of morbidities other than IA that may explain reduced work ability.
* Is under examination for comorbidities that influence work ability.
* Major surgery was conducted within the past six months, or a surgery has been planned.
* Is unable to understand or speak Danish at a sufficient level to participate.
* Has cognitive or psychological impairments that may affect participation.
* Planned or ongoing participation in another rehabilitation program (apart from physiotherapy).
* Has participated in the WORK-ON feasibility study.
* Retirement application process is ongoing or plans to retire within the next five years.
* Has taken long-term sick leave (>4 weeks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Work Ability Index (WAI) single item | Baseline to 6 months after baseline
  A visual analogue scale that compares perceived work ability with lifetime best score. The score ranges from 0 (completely unable to work) to 10 (work ability at its best)

SECONDARY OUTCOMES:
Job loss | 6,12,18 and 30 months after baseline
  Number of participants who currently has a job
Work hours per week | Baseline, 6,12,18 and 30 months after baseline
  Number of work hours per week
Work Productivity and Activity Impairment questionnaire, general health (WPAI:GH) | Baseline, 6,12,18 and 30 months after baseline
  Measures Absenteeism, Presenteeism, Overall work impairment and Activity impairment.
Sickness absenteeism | Each month after baseline during the 6 month intervention period via text message reminders.
  Days and hours of sick leave
Work ability in relation to demands | Baseline, 6,12,18 and 30 months after baseline
  Work Ability Index (WAI), question 2 Includes two questions about current work ability in relation to physical and mental demands.
Job insecurity | Baseline, 6,12,18 and 30 months after baseline
  Work ability Index (WAI) question 6 Do you believe, according to your present state of health, that you will be able to do your current job two years from now?"
Physical activity while at work | Baseline, 6 and 12 months after baseline
  Standing or walking with lifting or carrying Physically demanding job Mostly stationary work Mostly standing or walking
Occupational balance | Baseline, 6 and 12 months after baseline
  Occupational Balance Questionnaire (OBQ-11) that measures measures the participant's experience of balance in the amount and variation of their everyday activities.
Health related quality of life | Baseline, 6 and 12 months after baseline
  EuroQol-5 Dimensions, 5 levels (EQ-5D-5L) is a generic measure to assess population health. Includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) -1 to 1, worst to best.
VAS Pain | Baseline, 6 and 12 months after baseline
  Visual analogue scale (VAS) pain, measuring self-rated pain at the moment from 0-10 One question encompassing pain experienced over the previous four weeks and to what extent physical pain affected work and household chores
Fatigue | Baseline, 6 and 12 months after baseline
  Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales version 2 (BRAF-NRSv2) is three separate numerical rating scales (scored from 0-10, higher is better), which cover three items: fatigue level (severity), effect on life (impact), and coping
Physical activity | Baseline, 6 and 12 months after baseline
  Over the previous year, how would you describe your physical activity? How many days a week are you physically active for at least 30 minutes?
Mental well-being | Baseline, 6 and 12 months after baseline
  WHO-5 Well-being Index, The 5-item Well-Being Index is a generic rating scale measuring subjective well-being.
Sleep | Baseline, 6 and 12 months after baseline
  Number of hours and minutes of sleep during a normal night the previous 4 weeks During the previous 4 weeks, did you get enough sleep to feel rested?
  Questions about how you sleep:
  Did you have trouble falling asleep? Did you wake up several times at night and have difficulty falling asleep? Did you wake up early and were unable to fall asleep again? Did you sleep restlessly?
Work Ability Index (WAI) single item | 12, 18 and 30 months after baseline
  A visual analogue scale that compares perceived work ability with lifetime best score (0-10) The score ranges from 0 (completely unable to work) to 10 (work ability at its best)

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Hospital for Rheumatic Diseases, Sønderborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to the General Data Protection Regulations and Danish law on data protection we are not allowed to make IPD available to other researchers

REFERENCES:
- [Derived] Madsen CMT, Primdahl J, Christensen JR. Testing the efficacy of WORK-ON: vocational rehabilitation for people with chronic inflammatory arthritis in Denmark-protocol for a randomised controlled trial. BMJ Open. 2024 Nov 27;14(11):e089050. doi: 10.1136/bmjopen-2024-089050. PMID 39609020